CLINICAL TRIAL: NCT06375564
Title: An Open-Label, Non-Randomized, Single-Center, Investigator-Initiated Trial to Determine the Effectiveness of 177Lu-AB-3PRGD2 in Various Solid Tumors With Integrin αvβ3 Positive Expression
Brief Title: Clinical Evaluation of 177Lu-AB-3PRGD2 in Various Solid Tumors With Integrin αvβ3 Positive Expression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMYY-2020KY067-05
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-04

CONDITIONS: Refractory Solid Tumor
Keywords: Refractory Solid Tumor; Radioligand therapy; 177Lu-AB-3PRGD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-AB-3PRGD2 (Experimental): 177Lu-AB-3PRGD2 A maximum of 4 cycles of 80 mCi (2.96 GBq) 177Lu-AB-3PRGD2, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 4 cycles, every 6 weeks
  Interventions: Drug: 177Lu-AB-3PRGD2 radioligand therapy

INTERVENTIONS:
Drug: 177Lu-AB-3PRGD2 radioligand therapy — Radioligand therapy using 177Lu-AB-3PRGD2 80 mCi (2.96 GBq) will be performed 6-weekly. A maximum of 4 cycles will be administered.

SUMMARY:
This is an open-label, non-controlled, non-randomized study to assess the therapeutic efficacy of 177Lu-AB-3PRGD2 in patients with various solid tumors who will undergo radioligand therapy using 177Lu-AB-3PRGD.

DETAILED DESCRIPTION:
Integrin αvβ3 is highly expressed in some tumor cells and neovascularization, which is an ideal target for diagnosis and treatment of solid tumors. 177Lu-AB-3PRGD2, is a kind of new drug based on independent research and development in China, providing an effective target for the treatment of tumors. All patients underwent whole-body 68Ga-RGD PET/CT for selection and accepted intravenous injection with a fixed dose of 2.96 GBq (80 mCi) of 177Lu-AB-3PRGD2 within one week. Treatment is planned for up to 4 cycles, and the time interval between cycles is 6 weeks. The primary endpoint assessed the preliminary treatment efficacy of 177Lu-AB-3PRGD2 used for radioligand therapy in patients with various advanced tumors. The secondary endpoint evaluates the safety of 177Lu-AB-3PRGD2.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Age 18 and older.
3. Confirmed unresectable or metastatic refractory cancer with measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis).
4. Progressive disease after multiple-lines treatment.
5. Eastern Cooperative Oncology Group Performance Status ≤ 3.
6. Participant must have completed prior therapy at least 2 weeks (washout period) before 68Ga-RGD PET/CT scan. Any clinically significant toxicity (with the exceptions of hair loss and sensory neuropathy) related to prior therapy resolved below Grade 2 or baseline. Completion of entry into 68Ga-RGD study and completion of the scan.
7. Hematologic parameters are defined as Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 Platelet count ≥ 50,000/mm3 Hemoglobin ≥ 8 g/dL.
8. Blood chemistry levels defined as AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN) Total bilirubin ≤ 3 times ULN Creatinine ≤ 3 times ULN Able to remain motionless for up to 30-60 minutes per scan.

Exclusion Criteria:

1. Participant on any chemical anticoagulant including antiplatelet agents (excluding ASA).
2. Participants with Class 3 or 4 NYHA Congestive Heart Failure.
3. Clinically significant bleeding within two weeks before trial entry (e.g. gastrointestinal bleeding, intracranial bleeding).
4. Pregnant or lactating women.
5. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e. larger than what is required for placement of a central venous access, percutaneous feeding tube, or biopsy) within 28 days before study day 1 or anticipated surgery within the subsequent 6 weeks.
6. Has an additional active malignancy requiring therapy within the past 2 years.
7. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
8. Psychiatric illness/social situations that would interfere with compliance with study requirements
9. Cannot undergo PET/CT scanning because of weight limits (350 lbs).
10. INR>1.2; PTT>5 seconds above UNL.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of Cycle 4 (each cycle is 42 days)
  68Ga-RGD will be performed for efficacy evaluation by RECIST 1.1. Particularly, 68Ga-RGD will be performed at baseline, and 6 weeks after two treatment cycles.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events (safety and tolerability) | At the end of Cycle 4 (each cycle is 42 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. Dose-limiting toxicity was defined as any 177Lu-AB-3PRGD2-related AE ≥ grade 3 (G3). For Hemoglobin < 8.0 g/dL; < 4.9 mmol/L; < 80 g/L; Need blood transfusion heal. Severe hypocytosis or with this age group The total number of normal cells was reduced >50% and ≤75%.

CONTACTS AND LOCATIONS:
Overall Officials: Haojun Chen, MD, PhD, Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No